CLINICAL TRIAL: NCT04201301
Title: Knowledge, Attitude and Practice (KAP) for Egyptian Pediatric Dentists Regarding Usage of Stainless Steel Crown on Primary Molars Using Hall Technique: A Cross Sectional Study
Brief Title: Usage of Stainless Steel Crown on Primary Molars Using Hall Technique
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud mohamed El shafie, Principal Investigator, Cairo University
Other Study IDs: metal Crown and primary molars
Record Dates: First submitted 2019-12-12; First posted 2019-12-17 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rationale: Gaining information about the knowledge, practice and attitude regarding hall technique and find out how much the Egyptian dentists use this method for treatment the carious primary teeth.

Aim of the study: To assess the knowledge, practice and attitude of Egyptian dentists regarding non invasive restorative approach.

DETAILED DESCRIPTION:
The first study on the Hall Technique was published in 2006 . It was a retrospective study which analysed the practice records of a general dental practitioner from Scotland, Dr. Norna Hall. Dr. Hall simplified the standard technique to restore primary teeth using preformed SSCs and used it with her patients. This retrospective study involved a total of 978 crowns fitted in 259 children using her novel technique (today known as the Hall Technique). Most crowns were placed when there was clinical evidence of a proximal carious lesion into dentine and marginal ridge breakdown. This study showed the Hall Technique to have comparable outcomes to those achieved with other more conventional restorations.

Since then, growing understanding that caries is essentially a biofilm driven disease rather than an infectious disease, explains why the Hall Technique, and other 'sealing in' carious lesion techniques, are successful. The intervening ten years has seen robust evidence from several randomised control trials that are either completed or underway. These have found the Hall Technique superior to comparator treatments, with success rates (no pain or infection) of 99% (UK study) and 100% (Germany) at one year, 98% and 93% over two years (UK and Germany) and 97% over five years (UK). The Hall Technique is now regarded as one of several biological management options for carious lesions in primary molars.

ELIGIBILITY:
Inclusion Criteria:

1. Egyptian dentists.
2. Pediatric dentists ( having PhD).
3. Pediatric dentists (having Master degree or studying master degree) .

Exclusion Criteria:

1. dentists in other dental speciality.
2. dental students.
3. pediatric dentists who have not enough knowledge about hall technique.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Egyptian Paediatric in Hospitals and health care units
Sampling Method: Non-Probability Sample
Enrollment: 164 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
knowledge, practice and attitude of Egyptian Dentists regarding The Hall techniqu | baseline
  Measuring device: KAP Questionnare Measuring unit: Binary(Yes,No) + Multiple Choice Questions (MCQ).

CONTACTS AND LOCATIONS:
Overall Officials: faculty of dentistry cairo university, college, Study Director — Cairo University

REFERENCES:
- [Background] Innes NP, Evans DJ, Bonifacio CC, Geneser M, Hesse D, Heimer M, Kanellis M, Machiulskiene V, Narbutaite J, Olegario IC, Owais A, Araujo MP, Raggio DP, Splieth C, van Amerongen E, Weber-Gasparoni K, Santamaria RM. The Hall Technique 10 years on: Questions and answers. Br Dent J. 2017 Mar 24;222(6):478-483. doi: 10.1038/sj.bdj.2017.273. PMID 28336976
- [Background] Santamaria R, Innes N. Sealing Carious Tissue in Primary Teeth Using Crowns: The Hall Technique. Monogr Oral Sci. 2018;27:113-123. doi: 10.1159/000487835. Epub 2018 May 24. PMID 29794469
- [Result] Roberts A, McKay A, Albadri S. The use of Hall technique preformed metal crowns by specialist paediatric dentists in the UK. Br Dent J. 2018 Jan 12;224(1):48-52. doi: 10.1038/sj.bdj.2018.4. PMID 29326453